CLINICAL TRIAL: NCT03087838
Title: Postoperative Delirium in Adult Patients After Elective Craniotomy Under General Anaesthesia: a Prospective Cohort Study
Brief Title: Postoperative Delirium in Adult Patients After Elective Craniotomy Under General Anaesthesia
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, professor, Capital Medical University
Other Study IDs: KY2017-018-02
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Intensive Care; Surgical; Postoperative Care; Neurosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- delirium group: CAM-ICU is positive within the first 24 hours after operation
- non-delirium group: CAM-ICU is negative within the first 24 hours after operation

SUMMARY:
Postoperative delirium may result in many adverse complications. At present little is known about postoperative delirium in patients after crniotomy because they may manifest similar symptoms to definitely delirium for some structural brain disease. Objective of this study is to find out incidence and risk factors of postoperative delirium in patients after elective craniotomy and also the relationship of postoperative delirium with clinical outcome.

DETAILED DESCRIPTION:
The study is a prospective single-center cohort study. Consecutive adult patients admitted to the ICU after elective craniotomy is enrolled. Richmond Agitation Sedation Scale (RASS) is used to assess level of consciousness of patients; if conditions met "RASS≥-3", the Confusion Assessment Method for the Intensive Care Unit will proceed to evaluate delirium signs in patients. Delirium is assessed every 12-hour shift within 3 days during the patient's ICU stay and ended when discharged from ICU or dead, time started at 9am and 9pm. On the third day after operation when most patients have been transferred to general ward, delirium was assessed only at 9am for follow-up studies. Patients is divided into two groups via assessment of CAM-ICU: delirium groups and non-delirium groups. Factors potentially related to postoperative delirium are collected and categorized as preoperative, intraoperative and postoperative in chronological order. Univariate analyses between delirium groups and non-delirium groups is performed. The stepwise backward logistic regression is carried out to identify the independent predictors of delirium. Patients will be followed up until hospital discharge, death or 90 days after the enrollment. Clinical outcome such as days on the mechanical ventilator, endotracheal extubation time, need for re-intubation and tracheotomy, unexpected reoperation within 72 h after surgery, length of stay in the ICU , hospital costs and mortality will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients after elective craniotomy under general anaesthesia and admitted to the ICU directly after surgery.

Exclusion Criteria:

1. Patients younger than 18 years
2. Patients with emergency operation
3. Patients with preoperative impairment of consciousness (GCS<8)
4. Patients with a past medical history of delirium or schizophrenia(evaluated by the medical document)
5. Patients withventriculoperitoneal shunt or endoscope operation
6. Patients with inability to communicate in the preoperative period(including language barrier)
7. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients After Elective Craniotomy Under General Anaesthesia
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | Within the first 24 hours after operation
  CAM-ICU is positive

CONTACTS AND LOCATIONS:
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Zhang G, Wang Y, Huang H, Li H, Li M, Yang C, Li M, Chen H, Jing B, Lin S. Alteration of default mode network: association with executive dysfunction in frontal glioma patients. J Neurosurg. 2022 Oct 14;138(6):1512-1521. doi: 10.3171/2022.8.JNS22591. Print 2023 Jun 1. PMID 36242576
- [Derived] Wang CM, Huang HW, Wang YM, He X, Sun XM, Zhou YM, Zhang GB, Gu HQ, Zhou JX. Incidence and risk factors of postoperative delirium in patients admitted to the ICU after elective intracranial surgery: A prospective cohort study. Eur J Anaesthesiol. 2020 Jan;37(1):14-24. doi: 10.1097/EJA.0000000000001074. PMID 31464712